CLINICAL TRIAL: NCT06200805
Title: A Study on the Intervention Effect of Tai Chi on College Students With Insomnia and the Potential Role of Inflammatory Factors
Brief Title: ai Chi Reduces Insomnia in College Students: Exploring Inflammatory Factor Roles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Wu Hai Lan, Chief Researcher, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WLan
Record Dates: First submitted 2023-12-09; First posted 2024-01-11 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Students With Sleep Disorders
MeSH Terms: interventions — Tai Ji

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Intensity Taijiquan Exercise Group (Experimental): 60 minutes of tai chi exercise 5 times a week
  Interventions: Behavioral: tai ji quan
- Moderate Intensity Taijiquan Exercise Group (Experimental): 60 minutes of tai chi exercise 3 times a week
  Interventions: Behavioral: tai ji quan
- control subjects (No Intervention): The control group did not implement any intervention and maintained a normal life and study status.

INTERVENTIONS:
Behavioral: tai ji quan — 24-Style Taijiquan as an Intervention for College Students with Insomnia
  Arms: High Intensity Taijiquan Exercise Group; Moderate Intensity Taijiquan Exercise Group

SUMMARY:
College student volunteers were recruited from a university in Anhui Province, China, and screened by the Pittsburgh sleep quality index (PSQI) scale, and those with PSQI scores higher than 7 were considered to have clinical insomnia, and insomniac college students screened were subjected to a 24-week 24-form taijiquan intervention, and the rest of the insomniac volunteers were randomly divided into the fast-walking group and the control group. As the most common form of physical exercise for college students and the easiest aerobic exercise, brisk walking was chosen as an intervention for insomniac college students to better compare the efficacy of tai chi with that of general aerobic exercise for insomnia. The taijiquan group performed taijiquan exercise three times a week for 60 minutes each time, the brisk walking group performed brisk walking training three times a week for 60 minutes each time, and the control group did not carry out any intervention and maintained a normal life and study status. Before the intervention, questionnaires were filled out and fasting elbow venous blood was drawn, and the staff uniformly explained the intervention-related contents and precautions, and after 24 weeks of intervention, the post-test questionnaires and fasting venous blood were filled out centrally.

DETAILED DESCRIPTION:
Insomnia: measured by PSQI scale. The scale was developed by Buysse et al, a neurologist at the University of Pittsburgh, USA, and has an overall internal consistency Cronbach's ɑ coefficient of 0.83.The scale was used to assess the quality of sleep of an individual in the last month, and consists of 19 self-assessed and 5 other-assessed entries, for a total of 24 items, where the 19th entry and the five other-assessed entries do not participate in the scoring. The 18 scoring items include seven dimensions: subjective sleep quality, time to sleep, sleep efficiency, sleep disorders, hypnotic drug use, and daytime functioning. Each dimension is scored on a scale of 0-3, and the cumulative score is the total PSQI score, which ranges from 0-21, with higher scores indicating poorer sleep quality, and PSQI scores greater than 7 are considered clinical insomnia.

Physical activity: was measured using the Physical activity rating scale-3 (PARS-3). The scale has a revised by Liang Deqing et al. with a retest reliability of 0.82. The scale determines the amount of exercise in terms of intensity, time, and frequency of participation in physical activities. Exercise volume = exercise intensity × time × frequency, intensity and frequency are scored on a scale of 1 to 5, assigning 1 to 5 points respectively, and time is scored on a scale of 1 to 5, assigning 0 to 4 points respectively. The score range of the scale was 0-100 points, and the score of ≤19 points was low exercise, 20-42 points was medium exercise, and ≥43 points was high exercise.

ELIGIBILITY:
Inclusion Criteria:

* Meet the diagnostic criteria of insomnia i.e. PSQI score ≥ 7;

  * Age between 18 and 25 years old; ③ Exercise of the study subjects is low exercise i.e. PARS-3 score ≤ 19;

    * Have not received any psychological and pharmacological treatments in the past one year;

      * Have no visceral diseases, normal vision and hearing; ⑥ Have good physical fitness and can perform basic intensity of physical exercise; ⑦ Have signed the informed consent form.

Exclusion Criteria:

* Recent cardiovascular disease, musculoskeletal disease and other diseases that affect normal sports training;

  * Serious mental illness; ③ Antibiotics within the past three months; ④ Serious autoimmune disease; ⑤ Those who refuse to participate in the research project.

Ages: 17 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-07-20 (Actual)

PRIMARY OUTCOMES:
Role effects of tai chi intervention in college students with insomnia | Minimum 12 weeks
  Insomnia: measured by PSQI scale. The scale was developed by Buysse et al, a neurologist at the University of Pittsburgh, USA, and has an overall internal consistency Cronbach's ɑ coefficient of 0.83.The scale was used to assess the quality of sleep of an individual in the last month, and consists of 19 self-assessed and 5 other-assessed entries, for a total of 24 items, where the 19th entry and the five other-assessed entries do not participate in the scoring. The 18 scoring items include seven dimensions: subjective sleep quality, time to sleep, sleep efficiency, sleep disorders, hypnotic drug use, and daytime functioning. Each dimension is scored on a scale of 0-3, and the cumulative score is the total PSQI score, which ranges from 0-21, with higher scores indicating poorer sleep quality, and PSQI scores greater than 7 are considered clinical insomnia.
  Use of this scale to assess the improvement of insomnia in insomniac college students using taijiquan
Changes in inflammatory factors before and after tai chi intervention | Minimum 12 weeks
  Fasting elbow vein blood of 2 ml was collected from college students in the tai chi group, the fast walking group, and the control group. 2 ml of blood was tested using Luminex multifactor assay technology. The levels of IL-2, IL-4, IL-6, IL-10, TNF-ɑ, IFN-Y, IL-8, IL-13, and IL-1 in the supernatant were measured.
  Inflammatory factor data before and after exercise were analyzed in each group to observe the level of inflammatory factor changes before and after taijiquan intervention and to explore the role played by inflammatory factor changes in taijiquan intervention for insomniac college students.

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China